CLINICAL TRIAL: NCT03154970
Title: Cervical Stabilization in Individuals With Obstructive Sleep Apnea: a Randomized Clinical Trial
Brief Title: Cervical Stabilization in Individuals With Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Santa Maria (Other)
Responsible Party: Principal Investigator, Eliane Correa, Professor, Universidade Federal de Santa Maria
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UFSM-AOS-01
Record Dates: First submitted 2017-05-07; First posted 2017-05-16 (Actual); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Obstructive Sleep Apnea
Keywords: Physical Therapy Specialty
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Obstructive sleep apnea group (G OSA) (Experimental): The cervical stabilization will be performed with craniocervical flexion training aiming to strength the deep cervical flexors. For this purpose a pressure biofeedback device (stabilizer) that allows progressive levels of pressure during exercise(22-30 mmHg) will be used, which will be increased according to the capacity of the individuals (avoiding compensations or pain). The participant will be instructed to perform the craniocervical flexion in the supine position, the duration of the contraction will be 10 seconds followed by 10 seconds of rest (3 sets of 10 repetitions). The sessions will be held 2 times in weeks, for 6 weeks.
  Interventions: Device: Craniocervical flexion training
- Control group (GC) (No Intervention): The GC will be reassessed after six weeks and the same G OSA treatment will be offered after this period.

INTERVENTIONS:
Device: Craniocervical flexion training — The cervical stabilization will be performed with craniocervical flexion training with two weekly sessions for 6 weeks
  Arms: Obstructive sleep apnea group (G OSA)

SUMMARY:
This study will be performed in people with obstructive sleep apnea, in which one group will receive treatment with cervical stabilization for six weeks and the control group will receive treatment after the interval of six weeks

DETAILED DESCRIPTION:
The objective of this study was to evaluate the muscle strength of the cervical flexor and extensor muscles, to investigate the presence of cervical dysfunction and temporomandibular dysfunction, as well as to verify the effects of cervical stabilization in individuals with obstructive sleep apnea (OSA). The research will be carried out at the Orofacial Motricity Laboratory of the Federal University of Santa Maria (UFSM) and the University Hospital of Santa Maria (HUSM). Men and women between 20 and 60 years of age with a diagnosis of OSA will be invited to participate in this study, confirmed by polysomnography. The sample will consist of 22 patients with OSA, 11 subjects in the OSA group (OSA G) and 11 in the control group (CG) randomly. At the initial evaluation, an anamnesis will be performed and participants will respond to the Epworth Sleepiness Scale (ESS), Pittsburgh Sleep Quality Index (PSQI) and STOP-Bang questionnaire. The craniocervical posture will also be evaluated through photogrammetry (SAPo); The presence and severity of temporomandibular dysfunction (TMD) by the instruments Diagnostic Criteria in Research for Temporomandibular Dysfunction (RDC / TMD) and Temporomandibular Index (TMT); The presence of cervical dysfunction by the Craniocervical Dysfunction Index (CCID); The pressure pain threshold and the strength of the cervical flexor and extensor muscles, by pressure algometry and dynamometry, respectively. The OSA G will be submitted to cervical stabilization using the pressure biofeedback device (Stabilizer) and, after six weeks will be reassessed by the same questionnaires and instruments of the initial evaluation. The CG after six weeks will be reevaluated and the same treatment protocol will be offered.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 20 to 60 years;
* Clinical diagnosis of obstructive apnea of mild, moderate or severe sleep through polysomnography following the apnea / hypopnea index.

Exclusion Criteria:

* Body Mass Index (BMI) greater than or equal to 35 kg / m2;
* Use of continuous positive airway pressure;
* Diagnosis of neurological or neuromuscular disease;
* History of craniocervical trauma;
* Be under physiotherapeutic or speech-language therapy for, respectively, craniocervical and orofacial motor dysfunction or have performed in the last three months;
* Being in use of intraoral orthodontic appliances, which produce mandibular advancement

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2017-07-30 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
Change of sleep quality | Baseline and 7 weeks
  Sleep quality will be assessed twice through the Pittsburgh sleep quality index (PSQI), composed of nine self-administered questions, with scores scattered on a scale of zero to three. The sum of the responses provided by the overall score, which ranges from zero to 21, where the higher the score, the worse the quality of sleep.

SECONDARY OUTCOMES:
Change of craniocervical dysfunction index | Baseline and 7 weeks
  The craniocervical dysfunction index evaluates the cervical function and is composed of five items: amplitude of cervical movements, presence of pain to cervical movement, presence of noises and blockages in the cervical joints, pain on the palpation of the cervical muscles and craniocervical posture. For each evaluated item three scores are possible (0, 1 or 5) and the volunteers can be classified into four categories according to the severity of the dysfunction: no dysfunction (0 points), mild dysfunction (1 to 4 points), moderate dysfunction (5 to 9 points) and severe (10 to 25 points)
Change of pressure pain threshold | Baseline and 7 weeks
  The pressure pain threshold will be evaluated by means of an analog algometer (Wagner Instruments). This appliance has a 1 cm rubber ferrule attached at its end, which will be positioned perpendicular to the muscular surface.
  For this, the participants will be seated in a chair, with the trunk upright, back fully supported, feet resting on the ground and hands resting on the lower limbs. The pressure pain threshold will be bilaterally assessed in the masseter (upper, middle and lower) and temporal (anterior, middle and posterior) muscles, submandibular region, posterior mandibular region, sternocleidomastoid, upper trapezius and suboccipital muscles. All points will be gradually pressed up to the intensity that the participant reports any pain intensity, this value being visualized on the equipment and recorded as pain threshold at pressure.
Change of presence and and severity of temporomandibular dysfunction (TMD) | Baseline and 7 weeks
  The instrument that will be used to evaluate presence of TMD is Diagnostic criteria in research for temporomandibular disorders (RDC / TMD), which is divided in 2 axis: in Axis I allows the measurement of TMD signs and symptoms (physical evaluation) and in Axis II it evaluates the psychological and psychosocial factors (questionnaire).
  To measure TMD severity the Temporomandibular Index (TMI) is used, this result is obtained from RDC/TMD data from Axis I. Result is a qualification among light (0 to 0,3), moderate (0,3 a 0,6) or severe (0,6 to1) TMD according to TMI calculated.
Change of cervical posture | Baseline and 7 weeks
  The posture of the head and cervical spine will be evaluated by means of digital photography, with posterior analysis in the Postural Evaluation Software (SAPo v 0.68®). The anatomical points of the tragus, spinous process of the seventh cervical vertebra and orbicular commissure will be demarcated with Styrofoam balls in the participant's body.
Change of muscle strength | Baseline and 7 weeks
  The evaluation of muscle strength of cervical flexors and extensors will be performed using a Microfet 2 manual dynamometer (Hoggan Health industries, West Jordan, USA). For the assessment of cervical flexors, the participant will be positioned in the supine position, knees extended, head and neck in neutral position. The manual dynamometer will be positioned in the midline of the frontal bone and will be held by the evaluator, while the participant performs the maximum voluntary isometric contraction of the cervical flexors.
  In order to evaluate the strength of the cervical extensors the participant will be positioned in the prone position, with the upper limbs next to the trunk. The manual dynamometer will be positioned in the line of the occipital protuberance.
  Data from three repetitions will be obtained for flexion and cervical extension, each repetition lasts 5 seconds and the rest period between the repetitions is 60 seconds.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal de Santa Maria, Santa Maria, Rio Grande do Sul, Brazil